CLINICAL TRIAL: NCT01317264
Title: β-Glucans and the Metabolic Syndrome - a Human Intervention Study Under BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Susanne Gjedsted Bügel, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: M196
Record Dates: First submitted 2011-03-11; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: β-glucan; cholesterol; bile acids; blood glucose; appetite

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo milk drink (Placebo Comparator)
  Interventions: Other: no β-glucan
- Millk drink with oat β-glucan (Experimental)
  Interventions: Other: oat β-glucan
- Milk drink with barley β-glucan (Experimental)
  Interventions: Other: barley β-glucan
- Milk drink with mutant-barley β-glucan (Experimental)
  Interventions: Other: mutant-barley β-glucan

INTERVENTIONS:
Other: no β-glucan — daily consumption of non-β-glucan containing milk drinks together with the 3 main meals for 21 days
  Arms: Placebo milk drink
Other: oat β-glucan — daily consumption of 5g of oat β-glucan in the form of milk drinks with the 3 main meals for 21 days
  Other Names: "PromOat",Biovelop, Kimstad, Sweden
  Arms: Millk drink with oat β-glucan
Other: barley β-glucan — daily consumption of 5g β-glucan extracted from the barley-mutant mother "Bomi" in the form of milk drinks with the 3 main meals for 21 days
  Arms: Milk drink with barley β-glucan
Other: mutant-barley β-glucan — daily consumption of 5g β-glucan extracted from the high β-glucan barely mutant "lys. 5.f" in the form of milk drinks with the 3 main meals for 21 days
  Arms: Milk drink with mutant-barley β-glucan

SUMMARY:
The aim of this study is to investigate the potential disease preventive effects of β-glucans from oat and barley.

DETAILED DESCRIPTION:
Objective:

The primary aim is to examine whether consumption of oat and two different barley β-glucans exhibits hypocholesterolemic effects and to understand the underlying mechanisms.

Secondary aims are to investigate whether there are also effects on blood pressure, appetite regulation, insulin sensitivity, hemostasis, low-grade inflammation and the metabolic profile of different biological materials.

Intervention:

In each of the 4 intervention periods the participants drink a milk drink together with their three main meals for 21 days. This way they consume 5g β-glucan/d form either oat or barley in the three treatment periods, otherwise they maintain their habitual diet. They are not, however, allowed to eat any oat- or barley-containing products during the trial.

At the beginning and at the end of each intervention period the participants' blood pressure is measured and a fasting blood sample is drawn.

Further they collect feces for 72 hours and urine for 24 hours before and at the end of each intervention period.

Before and at the end of each intervention period a 4-hour meal test is undertaken to measure their subject appetite sensation. Here at first a fasting blood samples drawn and thereafter the milk drink is served. Appetite sensation is assessed every 30 min for 4 hours. Also blood samples are drawn at 2 hours and 4 hours at the meal tests which takes place before each intervention period.

At the subsequent "ad libitum" lunch meal the food intake is measured and then a final appetite registration is made.

Furthermore participants make 4-d food records before and at the end of each intervention period.

ELIGIBILITY:
Inclusion Criteria:

* normal weight or moderately overweight (BMI 18.5-30 kg/m²)

Exclusion Criteria:

* chronic diseases (e.g. diabetes, cardiovascular disease)
* elevated blood pressure
* hyperlipidemia
* consumption of dietary supplements during or 2 month prior to start of study (including vitamin tablets)
* consumption of oat and barley products from January 1st until the end of study
* smoking
* excess physical activity (> 8h/week)
* medicine use (not included contraceptives or occasional pain killer consumption)
* pregnancy
* breast feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
change in total and LDL cholesterol concentration | fasting blood sample at baseline and day 21
pH, SCFA, bile acids, total fat, total energy, cholesterol (in 72h feces) | average over three days at baseline and after 3 weeks
weight | at baseline and after 1, 2 and 3 weeks
food intake (in 4d records) | at baseline and after 3 weeks
height | at baseline

SECONDARY OUTCOMES:
insulin, glucose, IL-6, CRP, TNF-α, fibrinogen, PAI-1, appetite regulation peptides, alkylresorcinol, metabolomics (in fasting and meal test blood samples) | fasting blood sample at baseline and on day 21
appetite sensation (in meal tests) | 3h appetite registrations at baseline and on day 21
metabolomics, isoprostanes (in 24h urine) | at baseline and after 3 weeks
metabolomics (in 72h feces) | average over 3 days at baseline and after 3 weeks
blood pressure | at baseline and on day 21

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Principal Investigator — Department of human nutrition, University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark